CLINICAL TRIAL: NCT06208735
Title: CLIC-02: A Phase I Trial of CLIC-2201 for the Treatment of Relapsed/Refractory B Cell Malignancies
Brief Title: CLIC-2201 for the Treatment of Relapsed/Refractory B Cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIC-02
Record Dates: First submitted 2023-12-20; First posted 2024-01-17 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: B-Cell Leukemia; Non-Hodgkin's Lymphoma; B-cell Acute Lymphoblastic Leukemia; Diffuse Large B Cell Lymphoma; High-grade B-cell Lymphoma; Primary Mediastinal Large B-cell Lymphoma (PMBCL); Mantle Cell Lymphoma; B-cell Lymphoma
Keywords: Chimeric Antigen Receptor T cells; CLIC-2201; CD22; Immunotherapy; CAR-T cell
MeSH Terms: conditions — Leukemia, B-Cell; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, B-Cell

STUDY DESIGN:
Intervention Model Description: This is a Phase I, first-in-human, open-label multicenter trial of CLIC-2201 CAR-T cells in participants with relapsed or refractory CD22-positive B-cell malignancies. The trial will consist of a 3+3 dose-escalation/de-escalation method in both cohorts (Cohort A: individuals who are 18 years or older and diagnosed with relapsed or refractory B-NHL and Cohort B: pediatric individuals who are 1-21 years old and diagnosed with relapsed or refractory B-ALL) to evaluate the safety and tolerability of increasing dose levels of CLIC-2201 in order to estimate the MTD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CLIC-2201 (Experimental): A single Intravenous infusion of CLIC-2201 will be given.
  Interventions: Biological: CLIC-2201

INTERVENTIONS:
Biological: CLIC-2201 — Participants will undergo (a) lymphodepletion with cyclophosphamide and fludarabine, followed by (b) infusion of autologous CLIC-2201 CAR-T cells. All treatments will be delivered intravenously.
  Other Names: Autologous CD22 targeting CAR-T cells

SUMMARY:
This is a phase I dose-finding trial of an autologous CD22 targeting chimeric antigen receptor (CAR)-T cell product, called CLIC-2201, for participants with relapsed/refractory B cell malignancies. In the proposed trial, eligible enrolled participants will undergo leukapheresis for autologous T cell collection to enable CLIC-2201 manufacturing, followed by lymphodepletion with cyclophosphamide and fludarabine, then intravenous infusion of the autologous CLIC-2201 product. The trial will use the 3+3 design to escalate or de-escalate the dose level of CLIC-2201 administered. Participants will be monitored for safety and tolerability up to day 365 following CLIC-2201 infusion.

The primary objective is to evaluate the safety and tolerability of CLIC-2201 and estimate the maximum tolerated dose (MTD) of CLIC-2201 in B-cell malignancies.

The secondary objectives are to evaluate the (i) feasibility; (ii) anti-tumour activity of CLIC-2201; (iii) and characterize the pharmacokinetic (PK) profile of CLIC-2201.

Exploratory objectives will include: i) characterizing the cellular and humoral immune responses against CLIC-2201 up to 1 year following infusion of CLIC-2201; (ii) characterizing the phenotype and gene expression profile of CLIC-2201 cells; (iii) evaluating immune and tumour cells at baseline and relapse for biomarkers of response or toxicity; (iv) evaluating serum cytokines, circulating tumour DNA (ctDNA) and B cell aplasia as biomarkers of clinical outcomes; and (v) assessing the quality of life.

DETAILED DESCRIPTION:
This is a Phase I, first-in-human, open-label multicenter trial of CLIC-2201 CAR-T cells for participants with relapsed/refractory B cell malignancies.

This trial will be conducted in two cohorts (cohort A, including 12 adult participants with B-NHL and cohort B, including 12 paediatric/young adult participants with B-ALL).

Consented participants will undergo a series of tests to confirm eligibility. Following eligibility confirmation, participants will undergo leukapheresis, which enables CLIC-2201 manufacturing. Leukapheresis is a procedure where white blood cells are collected from the blood. The collected cells will be shipped fresh to the Conconi Family Immunotherapy Laboratory (CFIL) in Victoria, BC, where manufacturing will take place.

At the CFIL lab, the autologous T cells will be selected, activated, and transduced with lentivirus to deliver the sdCD22 CAR transgene and then expanded over a period of 8 days in an automated, closed process on the CliniMACS Prodigy.

Participants will undergo lymphodepleting chemotherapy consisting of fludarabine (40 mg/m^2 daily x 3 days) and cyclophosphamide (500 mg/m^2 daily x 2 days) on trial days -4 and -3. The chemotherapy will deplete the exciting immune cells and give a chance to the infused CAR-T cells to expand and grow in the body.

Infusion of the autologous CLIC-2201 will follow at least 48 hours after but within seven days of completion of the last dose of fludarabine.

The standard 3+3 design will be used for CLIC-2201 administration to guide dosing and determination of the maximum tolerated dose (MTD). At each dose level, a decision will be made by the study team to escalate (E), stay at the current dose (S), de-escalate (D), or remove that dose level from further enrollment on trial (R) based on the number of dose-limiting toxicities (DLTs) evaluable participants who experience a DLT at that level.

There is no evidence that dosing of CAR-T cells/kg is different between paediatric and adult populations; however, most CAR-T cell products for B-ALL typically used a lower dose than for B-NHL. Therefore, in this trial, each dose level would start with the accrual of one adult participant in Cohort A before enrolling paediatric participants in Cohort B at that dose level. If a dose level is seen to be too toxic in Cohort A, this dose level will not be tested in Cohort B.

Participants in each cohort will be enrolled and treated in groups of n=3. The first 3 participants (group 1) will be treated at DL1. The first participant at this dose level will be staggered for a minimum of 28 days to allow for the full assessment of DLTs. After this, the other two participants enrolled at this level will be monitored for a minimum 14-day period. The staggered intervals pattern will be repeated for each dose level.

If none of the three participants in group 1 experiences a DLT, another group of three participants will be treated at the next higher dose level (DL2).

If >=2/3 participants experience a DLT, the dose will be de-escalated to DL-1, with de-escalation to DL-1 potentially occurring if both first 2 participants experience a DLT.

If 1/3 participants experience a DLT, an additional group of 3 more participants will be treated at the same dose level.

The dose escalation will continue until the maximum dose level (DL3) is reached without significant DLTs, or when at least 2/6 participants experience DLTs at a certain dose level (i.e., 33% of patients with a DLT at that dose level). The MTD will then be defined as the dose level just below this toxic dose level.

To receive the CLIC-2201 infusion, participants will be admitted to the in-patient unit, and they will remain at the hospital for a minimum of 7 days to be monitored closely for any complication, infection, and side effects. The participants will be discharged to the appropriate outpatient clinic if they are deemed medically stable after this time.

Participants will be seen at the outpatient clinic or daycare unit on days 10, 14, 21, 28, 60, 90, 180, and 365 after the CLIC-2201 infusion. They will continue with annual follow-up visits up to 15 years post-CLIC-2201 infusion.

ELIGIBILITY:
Inclusion Criteria in Cohort A:

Participants must meet the following criteria to be enrolled on the trial:

1. Participants in the cohort A must be 18 years of age or older of age at time of informed consent.
2. Participants must provide written informed consent. The investigator is responsible for obtaining written informed assent/consent for the subject after adequate explanation of the study design, anticipated benefits and the potential risks. Subjects should sign the most current REB approved assent/consent prior to any study specific activity or procedure is performed. (Sites will follow their REB board requirements for consenting).
3. Participants must have a relapsed or refractory B cell lymphoma, including one of the following:

   1. diffuse large B-cell lymphoma (DLBCL) not otherwise specified (NOS),
   2. high grade B cell lymphoma NOS,
   3. high grade B cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements,
   4. primary mediastinal large B-cell lymphoma (PMBCL),
   5. aggressive B cell lymphoma transformed from an indolent lymphoma,
   6. mantle cell lymphoma (MCL),
4. Participants must have refractory or relapsed disease, defined as one of the following:

   1. Relapse or refractory disease after at least 2 lines of therapy, OR
   2. Any relapse after autologous or allogeneic hematopoietic cell transplantation (HCT), OR
   3. Any relapse after CAR-T cell therapy.
5. Participants must have adequate organ function at enrolment, defined as:

   1. Left ventricular ejection fraction (LVEF) ≥40%,
   2. Creatinine clearance using Cockcroft-Gault of > 30 mL/min, AND
   3. ALP/ALT < 5X upper limit of normal (ULN), conjugated bilirubin < 2X ULN, and no evidence or history of liver cirrhosis.
6. Participants must have Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2 or Karnofsky Score ≥50%.
7. Females of child-bearing potential and sexually active males must agree to use a highly effective contraception method (see section 5.4) through to at least one year following administration of the CLIC-2201 product.
8. Participants with accessible disease, willingness to undergo a tumour biopsy at enrolment. For participants with a recent (within 3 months) tumor biopsy, access to the archival biopsy is acceptable.

Inclusion Criteria in Cohort B:

1. Participants in the cohort B must be between 1-21 years of age at the time of consent.
2. Parent or legal guardian of the participant signed the informed consent and the participant's assent/consent is obtained (if applicable). The investigator is responsible for obtaining written informed assent/consent for the subject or legally acceptable representative (e.g. parent, legal guardian) after adequate explanation of the study design, anticipated benefits and the potential risks. Subjects should sign the most current REB approved assent/consent prior to any study specific activity or procedure is performed. (Sites will follow their REB board requirements for consenting).
3. Participants must have a relapsed or refractory B cell acute lymphoblastic leukemia (B-ALL).
4. Participants must have refractory or relapsed disease, defined as one of the following:

   1. Relapse or refractory disease after at least 2 lines of therapy, OR
   2. Any relapse after autologous or allogeneic hematopoietic cell transplantation (HCT), OR
   3. Any relapse after CAR-T cell therapy.
5. Participants in cohort B and/or those who have received CD22 targeted therapy must have documentation of CD22 tumour expression within the 6 months prior to study screening, and after any prior CD22 directed therapy (if applicable).
6. Participants must have adequate organ function at enrolment, defined as:

   1. Left ventricular ejection fraction (LVEF) ≥45%,
   2. Creatinine clearance using Cockcroft-Gault or Schwartz equation of > 30 mL/min, AND
   3. ALP/ALT < 5X upper limit of normal (ULN), conjugated bilirubin < 2X ULN, and no evidence or history of liver cirrhosis.
7. Participants must have a Karnofsky or Lansky Score ≥50%.
8. Participants in reproductive age must agree to use a highly effective contraception method (see section 5.4) through to at least one year following administration of the CLIC-2201 product.
9. Participants willingness to undergo a bone marrow biopsy at enrolment.

Exclusion Criteria:

1. Any uncontrolled or serious active infection at the time of enrolment.
2. Active autoimmune disease requiring immunosuppressive therapy within 4 weeks of enrolment.
3. Live vaccine ≤6 weeks prior to enrolment
4. Active Graft Versus Host Disease (GVHD) requiring systemic immunosuppressive therapy within 4 weeks of enrolment.
5. Treatment with any of the following in the specified time period before leukapheresis:

   1. Allogeneic HCT within 3 months,
   2. Autologous HCT within 3 months,
   3. CD19 CAR-T cell infusion within 3 months,
   4. Donor lymphocyte infusion (DLI) within 3 months,
   5. Bendamustine within the last 6 months,
   6. Any investigational agent within 30 days or 5 half-lives (whichever is shorter),
   7. Systemic administration of therapeutic dose corticosteroids (>20 mg/day prednisone or equivalent for adults and ≥ 12 mg/m2/day for paediatric participants) within 7 days prior to leukapheresis.
   8. Immunosuppressive therapies (i.e., calcineurin inhibitors, methotrexate, mycophenolate, rapamycin) within 4 weeks.
   9. Oral chemotherapy agents (i.e., venetoclax) within 5 half-lives. An exception to this is that bruton tyrosine kinase (BTK) inhibitors like ibrutinib can be continued in participants with mantle cell lymphoma throughout the trial period.
6. Other concurrent malignancy or a prior malignancy treated within the past 2 years, except carcinoma in situ of the skin or cervix treated with curative intent and with no evidence of active disease.
7. Concomitant genetic syndrome associated with bone marrow failure such as Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure or immunodeficiency syndrome.
8. Active (confirmed by PCR) hepatitis B or hepatitis C at time of screening confirmed by PCR.
9. Any Human Immunodeficiency Virus (HIV) infection at time of screening.
10. Hypersensitivity to fludarabine or cyclophosphamide.
11. Any allergy to gentamycin or its derivatives
12. Pregnant or nursing participants.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Defining the maximum tolerated dose (MTD) of CLIC-2201 | Within the first 28 days of CAR-T infusion
  The MTD will be measured by monitoring and recording the AEs experienced by the participant within the first 28 days after the infusion, including the treatment-related death as deemed by the investigator, grade 3 Cytokine Release Syndrome (CRS), Immune Effector Cell Associated Neurotoxicity Syndrome (ICANS), and Immune Effector Cell-Associated Hemophagocytic Lymphocytosis-Like Syndrome (IEC-HS) lasting for more than seven days; grade 4 CRS, ICANS, and IEC-HS; grade 4 non-hematologic toxicity that is not deemed related to CRS, ICANS, IEC-HS (except for Grade 4 transaminases and isolated, asymptomatic laboratory electrolyte abnormalities for seven days or more).
Proportion of participants who experienced any grade of CRS to define the safety of CLIC-2201 | Within the first 28 days of CAR-T infusion
  The safety will be measured by the proportion of participants who experienced any grade of CRS, ICANS, IEC-HS, any adverse events, and any severe adverse events.
Proportion of participants who experienced any grade of ICANs to define the safety of CLIC-2201 | Within the first 28 days of CAR-T infusion
  The safety will be measured by the proportion of participants who experienced any grade of CRS, any grade of ICANS, any adverse events, and any severe adverse events.
Proportion of participants who experienced any grade of IEC-HS to define the safety of CLIC-2201 | Within the first 28 days of CAR-T infusion
  The safety will be measured by the proportion of participants who experienced any grade of CRS, any grade of ICANS, any adverse events, and any severe adverse events.
Proportion of participants who experienced any grade of AEs to define the safety of CLIC-2201 | Within the first 28 days of CAR-T infusion
  The safety will be measured by the proportion of participants who experienced any grade of CRS, any grade of ICANS, any adverse events, and any severe adverse events.
Proportion of participants who experienced any SAEs to define the safety of CLIC-2201 | Within the first 28 days of CAR-T infusion
  The safety will be measured by the proportion of participants who experienced any grade of CRS, any grade of ICANS, any adverse events, and any severe adverse events.

SECONDARY OUTCOMES:
Proportion of participants achieving achieving and/or maintaining Complete response (CR) or complete response with incomplete count recovery (CRi). | Within 365 days of CAR-T infusion
  This would be used to measure the anti-tumour activities of the CLIC-2201 treatment within a year after the infusion. The complete response will be assessed on days 28, 90, 180, and 365.
  Response for lymphoma participants will be defined by Lugano criteria and for B-ALL participants by CIBMTR response criteria.
Proportion of participants with an overall response [achieving a CR or partial remission (PR)] | Within 365 days of CAR-T infusion
  This would be used to measure the anti-tumour activities of the CLIC-2201 treatment within a year after the infusion.
Proportion of B-ALL participants with B with minimal residual disease (MRD) negative status by next-generation sequencing and/or high-resolution flow cytometry. | Within 365 days of CAR-T infusion
  This would be used to measure the anti-tumour activities of the CLIC-2201 treatment within a year after the infusion. The partial remission will be assessed on days 28, 90, 180, and 365.
Overall survival rate | Up to 15 years of CAR-T infusion
  This would be used to measure the the anti-tumor activities of the CLIC-2201 treatment within 6 months after the infusion.
Progression free survival rate | Up to 15 years of CAR-T infusion
  This would be used to measure the the anti-tumor activities of the CLIC-2201 treatment within 6 months after the infusion.
The average number of CAR transgene copies per cell | Up to day 365
  This would be used to evaluate the pharmacokinetics of the CLIC-2201 treatment.
Proportion of participants who fail enrollment that were successfully screened | Enrollment
  This would be used to evaluate the feasibility of administering CLIC-2201 cells to participants with relapsed/refractory B Cell Malignancies.
Proportion of participants for whom leukapheresis failed that successfully completed trial enrollment | From date of enrollment until the date of leukapheresis, assessed up to 4 weeks
  This would be used to evaluate the feasibility of administering CLIC-2201 cells to participants with relapsed/refractory B Cell Malignancies.
Proportion of participants for whom CLIC-2201 manufacturing was unsuccessful that completed leukapheresis | Through manufacturing, an average of 8 days
  This would be used to evaluate the feasibility of administering CLIC-2201 cells to participants with relapsed/refractory B Cell Malignancies.
Proportion of participants who fail to receive CLIC-2201 infusion for whom a CLIC-2201 was successfully manufactured | Day of CLIC-2201 infusion
  This would be used to evaluate the feasibility of administering CLIC-2201 cells to participants with relapsed/refractory B Cell Malignancies.
Median time from enrollment to leukapheresis | From date of enrollment until the date of leukapheresis, assessed up to 4 weeks
  This would be used to evaluate the feasibility of administering CLIC-2201 cells to participants with relapsed/refractory B Cell Malignancies.
Median time from enrollment to CLIC-2201 infusion | From date of enrollment until the date of infusion, assessed up to 6 weeks
  This would be used to evaluate the feasibility of administering CLIC-2201 cells to participants with relapsed/refractory B Cell Malignancies.
Median time from enrollment to disease progression that prevents CLIC-2201 infusion. | From date of enrollment until the date of infusion, assessed up to 6 weeks
  This would be used to evaluate the feasibility of administering CLIC-2201 cells to participants with relapsed/refractory B Cell Malignancies.

OTHER OUTCOMES:
Serum cytokine levels before and after CAR-T cell infusion (Mesoscale) | Up to day 28 after the infusion
  This would be used to evaluate the biomarkers of CLIC-2201 treatment within 28 days after the infusion.
Proportion of participants with B-cell aplasia assessed by flow cytometry (BTNK panel) | Within 365 days after the infusion
  This would be used to evaluate the biomarkers of CLIC-2201 treatment within a year after the infusion. This would be assessed on days 28, 60, 90, 180, and 365.
Measurement (quantitative and qualitative) of circulating tumour DNA in peripheral blood. | Within 365 days after the infusion
  This would be used to evaluate the biomarkers of CLIC-2201 treatment within a year after the infusion.
Molecular profiling of tumour tissue to explore mechanisms of efficacy and resistance prior to CLIC-2201 infusion and on relapse. | At the time of enrollment and if relapsed (assessed up to 1 year post infusion)
  This would be used to evaluate immune and tumour cells at baseline and relapse for biomarkers of response or toxicity of CLIC-2201 treatment.
Total CD3, CD4 and CD8 absolute numbers and relative percentages (BTNK panel) | Up to 365 days after the infusion
  This would be used to evaluate immune and tumour cells at baseline and relapse for biomarkers of response or toxicity of CLIC-2201 treatment.
Phenotypic analysis of CLIC-2201 infusion product and cells in peripheral blood after CLIC-2201 infusion, as assessed by flow cytometry | Within 4 hours prior to infusion
  This would be used to characterize the phenotype and gene expression profile of CLIC-2201 cells.
Clonal typing and gene expression profiling of the CLIC-2201 infusion product. (Single cell RNA-sequencing) | Within 4 hours prior to infusion
  This would be used to to characterize the phenotype and gene expression profile of CLIC-2201 cells.
Evaluating the health-related quality of life | Up to 365 days after the infusion
  In Cohort A: EuroQol 5 Dimension 5 Level (EQ-5D-5L) will assess participants' quality of life across five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The questionnaire follows a five-level ranking system that ranges from no problems to extreme problems.
  In Cohort B:
  * For participants aged 16 or older: EQ-5D-5L will be used as above.
  * For participants aged 8 to 15: EQ-5D-Y will be used, which is the child-friendly version of the questionnaire above in five domains and a three-level ranking system that ranges from no problems to a lot of problems.
  * For participants aged 4 to 7, the proxy version of EQ-5D-Y will be used. In the proxy version, parent, caregiver, or informant will be asked to respond to the questionnaire by providing their own impression of participant's health status.
  * Participants aged 1 to 3 will not have a quality-of-life assessment.
Evaluating the quality of life | Up to 365 days after the infusion
  The EORTC Core Quality of Life questionnaire (EORTC C-30) will be used to assess physical, psychological, and social functions among participants in CLIC-2201 study. This questionnaire consists of 30 items organized into several multi-item scales and single-item measures.
  For the multi-item scale questions, the questionnaire uses a Likert scale format, with response options ranging from "Not at all" to "Very much," allowing patients to indicate the extent to which they have experienced each symptom or difficulty over the past week.
  The single-item questions focus on overall health and overall quality of life and the participants could circle a number between 1(very poor) to 7 (Excellent) to indicate how they felt during the past week.
Frequency of antibody responses against the single domain antibody (sdAb) portion of the CLIC-2201 CAR transgene | Within 365 days of CAR-T infusion
  This would be used to evaluate the immunogenicity of the CLIC-2201 treatment. This would be assessed on days 28, 90, 180, and 365.
Frequency of cellular immune responses against CLIC-2201 cells by ELISpot | Within 365 days of CAR-T infusion
  This would be used to evaluate the immunogenicity of the CLIC-2201 treatment. This would be assessed on days 28, 90, 180, and 365.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Hay, MD, Principal Investigator — BC Cancer
Locations (7):
- Canada (7):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Alberta Children's Hospital, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - BC Children's Hospital, Vancouver, British Columbia
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided